CLINICAL TRIAL: NCT05008666
Title: Induction Chemotherapy Sequential Sintilimab Combined With Dual Epigenetic Drugs (Chidamide and Azacitidine) in ENKTL-HLH: A Single-arm, Multi-center, Phase II, Exploratory Clinical Study
Brief Title: Induction Chemotherapy Sequential Sintilimab Combined With Dual Epigenetic Drugs for ENKTL-HLH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huiqiang Huang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELEN
Record Dates: First submitted 2021-08-14; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Safety and Efficacy
Keywords: sintilimab; chidamide; azacitidine; Extranodal NK/T cell lymphoma; hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphohistiocytosis, Hemophagocytic | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- L-DEP, Sintinimab+Chidamide, Sintinimab+Azacitidine (Experimental): 【L-DEP】
  L-asparaginase: 2000U/m2 d5, im
  Doxorubicin liposome: 25mg/m2 d1, ivd
  Etoposide: 100mg/m2 d1, d8, d15, ivd
  Methylprednisolone: 15mg/kg/day d1-3, 0.75mg/kg/day, d4-7, 0.25mg/kg/day, d8-14, ivd
  【Sintinimab+Chidamide】
  Sintinimab: 200mg，d1,ivd,q21d Chidamide：30mg biw, continued oral
  【Sintinimab+Azacitidine】
  Sintinimab:200mg，d1, ivd, q21d Azacitidine:75mg/m2, d1-d7, ih, q28d
  Interventions: Drug: Sintilimab; Drug: Chidamide; Drug: Azacitidine; Drug: L-DEP

INTERVENTIONS:
Drug: Sintilimab — 1. To evaluate the short-term objective efficacy of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  2. To evaluate the long-term efficacy and safety of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  3. Exploring biomarkers that may have predictive effects.
Drug: Chidamide — 1. To evaluate the short-term objective efficacy of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  2. To evaluate the long-term efficacy and safety of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  3. Exploring biomarkers that may have predictive effects.
Drug: Azacitidine — 1. To evaluate the short-term objective efficacy of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  2. To evaluate the long-term efficacy and safety of sintilimab Sequential combined with chidamide and azacitidine in the treatment of ENKTL-HLH patients.
  3. Exploring biomarkers that may have predictive effects.
Drug: L-DEP — L-DEP

SUMMARY:
ENKTL is a highly aggressive non-Hodgkin lymphoma closely related to EBV infection，and advanced patients often suffer from hemophagocytic lymphohistiocytosis (HLH). ENKTL-HLH lacks standard treatment and experiences a extremely poor prognosis. Anti-PD-1 antibody has shown good anti-tumor activity in ENKTL and play a potential role in EBV-HLH. Epigenetic drugs have been confirmed to exert synergistic anti-tumor activity with anti-PD-1 antibody. We next further explore the efficacy and safety of Sintilimab sequential combination of epigenetic drugs in ENKTL-HLH.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures.
2. The age at the time of signing the ICF is ≥18 years old and ≤75 years old.
3. ENKTL confirmed by the research center histopathology and HLH conformed by the HLH-2004 diagnostic criteria.
4. Available tumor tissue samples (10-15 unstained, fresh-frozen, paraffin-embedded [FFPE] glass slides) obtained from past or fresh coarse needle puncture or excision.
5. Newly treated or refractory or relapsed ENKTL that has failed treatment with asparaginase-based chemotherapy or radiochemotherapy.
6. HLH occurred for the first time.
7. Eastern cooperative oncology group score:0-2.
8. Estimated survival≥3 months.
9. There must be at least 1 evaluable or measurable lesion that meets the RECIL 2017 lymphoma standard [evaluable lesion: 18FDG/PET examination Shows increased local uptake in lymph nodes or extranodal areas (higher than liver) and PET and/or Computed Tomography (CT) features are consistent with lymphoma manifestations; measurable lesions: nodular lesions longer than 15mm or extranodal lesions longer diameter >10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of imaging progression after radiotherapy) and accompanied by increased 18FDG uptake]. No measurable lesion and the diffuse increased 18FDG uptake in the liver would be excluded.
10. Sufficient organ function, no serious heart, lung, kidney, thyroid dysfunction and immune deficiency:

    1. Hemoglobin ≥6 g/dL (no growth factor support or blood transfusion was used within 7 days before platelet measurement);
    2. Platelets ≥60×109/L (no growth factor support or blood transfusion was used within 7 days before platelet measurement);
    3. Serum creatinine ≤1.5 times the upper limit of normal (Upper Limit Normal, ULN), or creatinine clearance ≥40mL/min (estimated according to the Cockcroft-Gault formula);
    4. Serum total bilirubin ≤ 5 times ULN (unless it is confirmed to have Gilbert syndrome);
    5. Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) ≤10 times ULN;
    6. Coagulation function: International Normalized Ratio (INR)≤1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT)≤1.5 times ULN; Fiber Fibrinogen (Fbg)>1.0g/L. (Unless the subject is receiving anticoagulant therapy and PT and APTT are within the expected range of anticoagulant therapy at the time of screening).
    7. Thyroid stimulating hormone (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) are within ±10% of the normal value.
11. There is no evidence that the subject has difficulty breathing at rest, and the pulse oximetry value at rest is> 92%.
12. The subject must pass a pulmonary function test (PFT) to confirm that the forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is greater than 60%; the diffusion volume of carbon monoxide (DLCO), FEV1 and FVC are all exceeding the predicted value by 50 % Above; all PFT results must be obtained within 4 weeks before the first dose.
13. Subjects who have received anti-tumor therapy in the past should return to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 rating score ≤ level 1 or baseline level after the toxicity of the previous treatment has been restored Entry into the group; The irreversible grade 2 toxicity (such as thrombocytopenia, anemia, neurotoxicity, hair loss and hearing loss) caused by previous anti-tumor treatments and is not expected to worsen during the study treatment period requires the consent of the investigator to be included in the group.
14. Women of Childbearing Potential (WOBCP) must have a serum pregnancy test within 7 days before the first medication, and the result is negative; WOBCP or men and their WOBCP partners should agree from signing the ICF to the last dose Take effective contraceptive measures within 6 months after the study drug.

Exclusion Criteria:

1. Invasive natural killer cell leukemia.
2. Primary central nervous system lymphoma or secondary central nervous system involvement.
3. Have received other anti-tumor therapy (including chemotherapy, immunotherapy, targeted therapy, and allowed to receive L-DEP or HLH-94/04 regimen for HLH).
4. Have received allogeneic organ transplantation.
5. Received allogeneic hematopoietic stem cell transplantation (allo-HSCT) within 3 years before study drug administration (Patients who have received allo-HSCT more than 3 years before study drug administration and currently have no graft-versus-host reaction can be included in the group).
6. Participating in other clinical studies, or planning to start the treatment of this study is less than 4 weeks from the end of the previous clinical study.
7. An autologous hematopoietic stem cell transplantation(ASCT) was performed within 90 days.
8. Received immune checkpoint inhibitors (anti-PD-1/PD-L1/CTLA-4 antibodies and other drugs) within half a year.
9. Have received histone deacetylase inhibitor or DNA methyltransferase inhibitor treatment within 1 year before the study drug administration.
10. Suffer from active autoimmune diseases that require systemic treatment in the past two years (glucocorticoid replacement therapy is not considered systemic treatment, such as type I diabetes, hypothyroidism that requires only thyroxine replacement therapy, only Patients with low adrenal function or hypopituitarism who need to receive physiological doses of glucocorticoid replacement therapy); patients with autoimmune diseases who do not require systemic treatment in the past two years can be included in the group.
11. Subjects who need to receive systemic glucocorticoid therapy or other immunosuppressive therapy due to certain conditions within 14 days before starting the research treatment [Subjects are allowed to use topical, ocular, intra-articular, intranasal and inhaled types glucocorticoid therapy (very low systemic absorption); high-dose intravenous or oral glucocorticoid therapy for HLH is allowed; short-term (≤ 7 days) use of glucocorticoid for preventive treatment (such as contrast agent allergy) or for the treatment of non-autoimmune diseases (for example, delayed-type hypersensitivity reactions caused by contact allergens)].
12. Suffered from other malignant tumors in the past 5 years, except for skin basal cell carcinoma, skin squamous cell carcinoma, breast carcinoma in situ and cervical carcinoma in situ that have undergone radical treatment.
13. Received systemic anti-tumor therapy within 28 days before starting the study drug treatment, including chemotherapy, immunotherapy, biological therapy (tumor vaccine, cytokines, or growth factors), etc. [L-DEP or HLH-94/04 based regimens are allowed for HLH; G-CSF,IL-11, TPO, EPO therapy are allowed.
14. Received major surgery within 28 days or radiation therapy within 90 days.
15. Received traditional Chinese medicine or Chinese patent medicine treatment within 7 days.
16. Vaccine live vaccines (except influenza attenuated vaccine) within 28 days.
17. Human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome.
18. Patients with active chronic hepatitis B or active hepatitis C. In the screening period, patients who are positive for Hepatits B Surface Antigen (HBsAg) or Hepatitis C Virus (HCV) antibodies must pass the Hepatitis B Virus (HBV) DNA titer test (not allowed Higher than 2500 copies/mL or 500 IU/mL) and HCV RNA testing (not exceeding the lower limit of detection of the assay). After excluding the active hepatitis B or C infection that requires treatment, the test can be included . Carriers of hepatitis B virus, hepatitis B (DNA titer shall not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and hepatitis C patients who have been cured can be included in the group.
19. Active tuberculosis.
20. Active fungal, bacterial and/or viral infections that require systemic treatment.
21. Women who are pregnant or breastfeeding.
22. People with a history of alcohol or drug abuse.
23. Suffer from uncontrollable comorbid diseases, including but not limited to symptomatic congestive heart failure, acute and chronic liver failure, uncontrollable hypertension, unstable angina, active peptic ulcer or bleeding disorders.
24. A history of interstitial lung disease or non-infectious pneumonia within 3 months before the start of the study treatment. Subjects who have previously had drug-induced or radioactive non-infectious pneumonia but asymptomatic are allowed to join the group.
25. QTcF interval> 450 msec, unless it is secondary to bundle branch block.
26. People with a history of mental illness; those who are incapacitated or restricted.
27. According to the judgment of the investigator, the patient's basic condition may increase the risk of receiving study drug treatment, or cause confusion about the toxic reaction and its judgment.
28. The investigator assessed that the patient was not suitable for participating in the study due to other conditions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) after end of treatment | [Time Frame: up to 24 months]
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Complete response rate (CRR) after end of treatment | [Time Frame: up to 24 months]
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)
Partial response rate (PRR) after end of treatment | [Time Frame: up to 24 months]
  Assessed by the lymphoma response to immunomodulatory therapy criteria (LYRIC)

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | [Time Frame: Time Frame: up to 36 months]
  PFS is defined as the time from the treatment date to the date of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
Overall Survival (OS) | [Time Frame: up to 36 months]
  OS is defined as the time from treatment to the date of death.
Duration of Response (DOR) | [Time Frame: up to 36 months]
  Among participants who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the the lymphoma response to immunomodulatory therapy criteria (LYRIC) or death regardless of cause.
Time to disease response (TTR) | [Time Frame: up to 36 months]
  Among participants who experience an objective response, TTR is defined as the date of their first administration to the day of their first objective response (which is subsequently confirmed) per the RECIL 2017 Response Criteria for Malignant Lymphoma.
Time to progression (TTP) | [Time Frame: Up to 36 months]
  Among all participants, TTP is defined as the date of their first administration to the day of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
The frequency of adverse events (adverse events, AEs) and serious adverse events (SAEs) | [Time Frame: Up to 36 months]
  An adverse event (AE) is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAE were defined as AEs with onset during the treatment period or that are a consequence of a pre-existing condition that has worsened since baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology,Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided